CLINICAL TRIAL: NCT02511340
Title: Multi-center, Single Stage Phase II Study to Evaluate the Efficacy and Safety of Flumatinib in Accelerated or Blastic Phase Chronic Myelogenous Leukemia Patients
Brief Title: A Phase II Study to Evaluate the Efficacy and the Safety of Flumatinib in CML-AP or CML-BP Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HHGV678-204
Record Dates: First submitted 2015-07-26; First posted 2015-07-30 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Chronic Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Flumatinib mesylate tablet 600 mg qd (Experimental): Flumatinib, 600mg, qd
  Interventions: Drug: Flumatinib mesylate tablet 600 mg qd

INTERVENTIONS:
Drug: Flumatinib mesylate tablet 600 mg qd — Flumatinib mesylate tablet 600 mg qd in CML-AP or CML-BP patients

SUMMARY:
Multi-center, single stage, phase II study to evaluate the efficacy and safety of Flumatinib in accelerated or blastic Phase chronic myelogenous leukemia patients.

DETAILED DESCRIPTION:
Multi-center, single-arm, open-label,phase II study to investigate efficacy and safety of Flumatinib in Chinese patients with accelerated or blastic Phase chronic myelogenous leukemia. The starting daily oral dose of Flumatinib is 600mg，core test is six cycles (each cycle is 28 days), collecting the core test data for primary efficacy analysis. The longest treatment time is 12 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients age 18-75 year-old;
* ECOG 0 - 2;
* Newly diagnosed or previously treated Ph+ CML patients in accelerated or blastic Phase;
* Adequate organ function;
* Written informed consent prior to any study procedures being performed.

Exclusion Criteria:

* Patients in Chronic and Blastic Phases;
* Previously treated with Flumatinib;
* Previously documented T315I mutations;
* Previous therapy within protocol defined timeframe, including:

  * hydroxyurea within 24 hr,
  * Imatinib or Nilotinib or Dasatinib within 28 days)
* Cardiac dysfunction ;
* History of congenital or acquired bleeding disorders unrelated to CML;
* Central nervous system leukemia;
* Previous malignancy except CML;
* Acute or chronic liver or severe kidney disease unrelated to CML;
* Pregnant, breastfeeding, child bearing potential but failed to take effective contraception.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-08 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Confirmed overall hematologic response（OHR）at 6 months | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kaiyan Liu, Study Chair — Peking University People's Hospital
Locations (1):
- Union Hospital Tongji Medical College Huazhong University of Science and technology, Wuhan, Hubei, China